CLINICAL TRIAL: NCT05266820
Title: TACTIC: a Phase II Study of TAS-102 Monotherapy and Thalidomide Plus TAS-102 as Third-line Therapy and Beyond in Patients With Advanced Colorectal Carcinoma
Brief Title: Trifluridine/Tipiracil (TAS-102) With or Without Thalidomide for the Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTIC
Record Dates: First submitted 2022-01-13; First posted 2022-03-04 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Thalidomide; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAS-102+Thalidomide (Experimental): Thalidomide 100mg PO BID+TAS-102 35mg/m2, po, bid, d1-5, d8-12, q4wks
  Interventions: Drug: Thalidomide; Drug: TAS-102
- TAS-102 (Active Comparator): TAS-102 35mg/m2, po, bid, d1-5, d8-12, q4wks
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: Thalidomide — For the experimental group, the intervention was thalidomide（100mg PO Bid)
  Other Names: Thalidomide Tablets produced by Changzhou Pharmaceutical Factory Co. LTD
  Arms: TAS-102+Thalidomide
Drug: TAS-102 — TAS-102

SUMMARY:
Thalidomide has both anti-angiogenesis and antiemetic effects, and its combined use with TAS-102 may reduce the gastrointestinal reactions associated with TAS-102, while enhancing antitumor efficacy and reducing the side effects of chemotherapy, and its cost is significantly lower than that of bevacizumab, which has higher pharmacoeconomics and greater clinical research application value.

DETAILED DESCRIPTION:
In the past decade, the use of targeted drugs has greatly improved the overall survival of patients with mCRC. However, there are currently few effective drugs available clinically. Trifluridine/Tipiracil (TAS-102) is a novel cytotoxic antitumor drug taken orally with minor adverse reactions, consisting of trifluridine and tipyrimidine hydrochloride. Tas-102 has been approved for the treatment of patients with metastatic colorectal cancer (mCRC) who have been previously treated with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy; an anti-VEGF biological therapy; and if RAS wild type, an anti-EGFR therapy. Multiple studies have shown that TAS-102 prolongs median OS and PFS in mCRC patients compared with placebo.

Thalidomide is a sedative that was developed in the late 1950s and eventually marketed and prescribed in several countries to pregnant women to alleviate nausea in the late 1950s and early 1960s. The drug, however, caused severe birth defects in more than 10,000 children worldwide and was forced to withdraw from the international market. Further studies found that the S-optical isomer of thalidomide can inhibit neutrophil chemotaxis, produce anti-inflammatory activity, stimulate immune system activation, regulate immunity, anti-angiogenesis, and inhibit the adhesion of cancer cells to stroma, so as to change the microenvironment of the body, and achieve anti-tumor effect.

Thalidomide has both anti-angiogenesis and antiemetic effects, and its combined use with TAS-102 may reduce the gastrointestinal reactions associated with TAS-102, while enhancing antitumor efficacy and reducing the side effects of chemotherapy, and its cost is significantly lower than that of bevacizumab, which has higher pharmacoeconomics and greater clinical research application value.

ELIGIBILITY:
1. Have histological or cytological documentation of adenocarcinoma of the colon or rectum (mCRC).
2. For patients with disease progression after conventional treatment, TAS-102 is determined as the third-line therapy or beyond according to the routine treatment practice of the researcher.
3. Aged no less than 20 years.

5.Have a measurable disease, according to RECIST version 1.1 6.Eastern Cooperative Oncology Group performance status 0-2. 7.Life expectancy of at least 12 weeks. 8.For women with reproductive potential, serum tests were performed within 7 days before the start of study treatment β- Human chorionic gonadotropin (β- HCG) pregnancy test, the result is negative. Women with reproductive potential must agree to take appropriate contraceptive measures with informed consent until at least 6 months after the last use of the study drug.

9.Sufficient bone marrow, liver and kidney functions and meet the following laboratory requirements:

1. Platelet count ≥75 × 109 /L
2. Hemoglobin level ≥90 g/L
3. Absolute neutrophil count ≥1.5× 109 /L

a) Total bilirubin ≤1.5 × upper limit of normal (ULN) b) Alanine aminotransferase and aspartate aminotransferase ≤2.5 × ULN (≤5 × ULN for patients with liver metastases) d) Serum creatinine ≤1.5 × ULN e) Glomerular filtration rate ≥30 ml/min/1.73 m2, according to the modified diet in renal disease abbreviated formula 10.Able to take oral drugs. 11.Have signed written informed consent.

Exclusion criteria

1. With arterial or venous thrombosis or embolic events such as myocardial infarction, cerebral thrombosis, intracerebral hemorrhage, deep venous thrombosis or pulmonary embolism within 6 months before the start of the study.
2. Evidence or history of any bleeding diathesis, irrespective of severity. Any hemorrhage or bleeding event ≥ grade 3 (adverse events per CTCAE v5.0) within 4 weeks prior to the start of treatment.
3. Peripheral neuropathy > grade 1 (adverse events per CTCAE v5.0).
4. History of uncontrolled or medicated heart disease.
5. Seizure disorder requiring medication.
6. Known history of human immunodeficiency virus (HIV) infection.
7. Patients with an active infection.
8. Other uncontrolled concurrent diseases determined by the researchers as not meeting the study conditions.
9. Patients with ascites and pleural effusion with clinical symptoms requiring treatment.
10. Known allergy to any of the study drug ingredients.
11. Unable to swallow oral medication.
12. Prior exposure to TAS-102 or thalidomide.
13. Patients who have brain metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS was defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.

SECONDARY OUTCOMES:
Overall survival（OS） | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  OS was defined as the time from the date of randomization to the date of death due to any cause. For subjects who were alive or lost to follow-up by the data analysis cut-off date, survival was censored at the subject's last known survival time.
Incidence of Treatment-Emergent Adverse Events | from first dose to within 30 days after the last dose
  Incidence of Treatment-Emergent Adverse Events were evaluated in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Fujian Medical University Cancer Hospital, Fujian Cancer Hospital, Fuzhou, Fujian
  - First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Fujian Provincial people's Hospital, Fuzhou
  - Fuzhou First Hospital affiliated to Fujian Medical University, Fuzhou
  - Hospital 900 of the Joint Logistic Support Force of the Chinese People's Liberation Army, Fuzhou
  - The Third People's Hospital affiliated to Fujian University of Chinese Medicine, Fuzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Ma J, Yang QL, Ling Y. Rechallenge and maintenance therapy using cetuximab and chemotherapy administered to a patient with metastatic colorectal cancer. BMC Cancer. 2017 Feb 14;17(1):132. doi: 10.1186/s12885-017-3133-8. PMID 28196490
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Andersen SE, Andersen IB, Jensen BV, Pfeiffer P, Ota T, Larsen JS. A systematic review of observational studies of trifluridine/tipiracil (TAS-102) for metastatic colorectal cancer. Acta Oncol. 2019 Aug;58(8):1149-1157. doi: 10.1080/0284186X.2019.1605192. Epub 2019 Apr 19. PMID 31002008
- [Background] Wallander M, Rolander B, Avall-Lundqvist E, Elander NO. Real world aspects of palliative trifluridine plus tiperacil (TAS-102) in refractory metastatic colorectal cancer. J Gastrointest Oncol. 2020 Aug;11(4):616-625. doi: 10.21037/jgo-20-43. PMID 32953145
- [Background] Longo-Munoz F, Argiles G, Tabernero J, Cervantes A, Gravalos C, Pericay C, Gil-Calle S, Mizuguchi H, Carrato-Mena A, Limon ML, Garcia-Carbonero R. Efficacy of trifluridine and tipiracil (TAS-102) versus placebo, with supportive care, in a randomized, controlled trial of patients with metastatic colorectal cancer from Spain: results of a subgroup analysis of the phase 3 RECOURSE trial. Clin Transl Oncol. 2017 Feb;19(2):227-235. doi: 10.1007/s12094-016-1528-7. Epub 2016 Jul 21. PMID 27443414
- [Background] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050
- [Background] Yoshida Y, Yamada T, Matsuoka H, Sonoda H, Fukazawa A, Yoshida H, Ishida H, Hirata K, Hasegawa S, Sakamoto K, Otsuka T, Koda K. A Trial Protocol of Biweekly TAS-102 and Bevacizumab as Third-Line Chemotherapy for Advanced/Recurrent Colorectal Cancer: A Phase II Multicenter Clinical Trial (The TAS-CC4 Study). J Anus Rectum Colon. 2019 Jul 30;3(3):136-141. doi: 10.23922/jarc.2018-043. eCollection 2019. PMID 31583329
- [Background] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574
- [Background] Liu H, Ma Y, Xu HC, Huang LY, Zhai LY, Zhang XR. Updates on the Management of Ocular Vasculopathies with VEGF Inhibitor Conbercept. Curr Eye Res. 2020 Dec;45(12):1467-1476. doi: 10.1080/02713683.2020.1781193. Epub 2020 Jul 7. PMID 32631094
- [Background] Kotani D, Kuboki Y, Horasawa S, Kaneko A, Nakamura Y, Kawazoe A, Bando H, Taniguchi H, Shitara K, Kojima T, Tsuji A, Yoshino T. Retrospective cohort study of trifluridine/tipiracil (TAS-102) plus bevacizumab versus trifluridine/tipiracil monotherapy for metastatic colorectal cancer. BMC Cancer. 2019 Dec 27;19(1):1253. doi: 10.1186/s12885-019-6475-6. PMID 31881856
- [Background] Eriksson T, Bjorkman S, Roth B, Fyge A, Hoglund P. Enantiomers of thalidomide: blood distribution and the influence of serum albumin on chiral inversion and hydrolysis. Chirality. 1998;10(3):223-8. doi: 10.1002/(SICI)1520-636X(1998)10:33.0.CO;2-A. PMID 9499573
- [Background] Zhang L, Qu X, Teng Y, Shi J, Yu P, Sun T, Wang J, Zhu Z, Zhang X, Zhao M, Liu J, Jin B, Luo Y, Teng Z, Dong Y, Wen F, An Y, Yuan C, Chen T, Zhou L, Chen Y, Zhang J, Wang Z, Qu J, Jin F, Zhang J, Jin X, Xie X, Wang J, Man L, Fu L, Liu Y. Efficacy of Thalidomide in Preventing Delayed Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase III Trial (CLOG1302 study). J Clin Oncol. 2017 Nov 1;35(31):3558-3565. doi: 10.1200/JCO.2017.72.2538. Epub 2017 Aug 30. PMID 28854065
- [Background] Melchert M, List A. The thalidomide saga. Int J Biochem Cell Biol. 2007;39(7-8):1489-99. doi: 10.1016/j.biocel.2007.01.022. Epub 2007 Jan 30. PMID 17369076
- [Background] Chen C, Yu G, Xiao W, Xing M, Ni J, Wan R, Hu G. Thalidomide inhibits proliferation and epithelial-mesenchymal transition by modulating CD133 expression in pancreatic cancer cells. Oncol Lett. 2017 Dec;14(6):8206-8212. doi: 10.3892/ol.2017.7213. Epub 2017 Oct 18. PMID 29344263
- [Background] 中国临床肿瘤学会（CSCO）.抗肿瘤治疗相关恶心呕吐预防和治疗指南（M）.（2019.V1.0）